CLINICAL TRIAL: NCT03675958
Title: Immediate Effect of Johnstone's Pressure Splint Added to Stretching on the Spasticity of Elbow Flexors and Wrist in Cerebrovascular Disease (CVD).
Brief Title: Immediate Effect of Johnstone's Pressure Splint Added to Stretching on the Spasticity in Cerebrovascular Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Industrial de Santander (Other)
Responsible Party: Principal Investigator, María Juliana González Silva, Physiotherapist, Universidad Industrial de Santander
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UISantander
Record Dates: First submitted 2018-09-01; First posted 2018-09-18 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Spasticity as Sequela of Stroke
Keywords: H Reflex; Johnstone's Pressure Splint; Stretching; Functional Reach; Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: A randomized experimental study with two intervention groups will be performed. Control group (GS): Stretching and experimental group: (GJPS + S): Johnstone´s Pressure Splint plus Stretching.
Who Masked: Investigator
Masking Description: The evaluator does not know the assignment of the participants to the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GJPS + S (Experimental): Experimental group: (GJPS + S) : Application Johnstone´s Pressure Splint plus Stretching in in 4 different treatment postures.
  Interventions: Other: Johnstone's Pressure Splint; Other: Stretching
- GS (Active Comparator): Control group (GS): Just Stretching in 4 different treatment postures.
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Johnstone's Pressure Splint — the intervention consists in the application of two tools used for the treatment of spasticity post - CVD. Johnstone's Pressure Splint added Stretching
  Arms: GJPS + S
Other: Stretching — the intervention consists in the application of one tool used for the treatment of spasticity post - CVD. Just Stretching

SUMMARY:
TITLE: Immediate effect of Johnstone's Pressure Splint added to Stretching on the spasticity of elbow flexors and wrist in Cerebrovascular Disease (CVD).

INTRODUCTION: In the rehabilitation of the upper limb post-CVD to employed exercise modalities such as stretching (S) to control spasticity, improve mobility and functionality. Also it is used the Johnstone´s Pressure Splint (JPS), which exerts circumferential pressure and contribute to spastic pattern inhibition, sensory re-education and increased of the mobility.

OBJECTIVE: The aim of the study is to evaluate the immediate effect of JPS added to S on the spasticity of elbow flexors and wrist, the reflex excitability and the joint kinematics in Stroke.

MATERIALS AND METHODS: A randomized experimental study with two intervention groups will be performed. Control group (GS): Stretching and experimental group: (GJPS + S): JPS plus S. Measurement times: Before the intervention (T0) and immediately post- intervention (T1). The outcome variables are muscle tone of elbow, wrist and hand assessed with the Modified Ashworth Scale (MAS); H reflex of the Flexor Carpi Radialis muscle, latency (ms), duration (ms) and amplitude (mV) of the M and H waves, and the amplitude the Hmax / Mmax ratio (%). Shoulder, elbow and trunk angles (degrees), trunk displacement (cm) and duration (sec) of the Functional Reach Pattern (PAF) will be evaluated with the software Contemplas.

ANALYSIS: Descriptive statistics will be applied and Shapiro Wilk test to evaluate the normality of the variables. Intra-group differences will be assessed with the student t-test paired and intergroup with the student t-test unpaired or the sum of Wilcoxon rank according to the distribution of the variables.

EXPECTED RESULTS: Hypotheses and contributions to the scientific evidence on the immediate effect of the S and JPS will be generated, to support the JPS as a complement to the traditional treatment. The results will be socialized in an international scientific event and a publication will be submitted to an impact journal.

KEY WORDS: Spasticity, H Reflex, Johnstone's Pressure Splint, Stretching, Functional Reach.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of CVD.
* Minimum evolution time from 6 months to 48 months.
* Muscular tone according to the Modified Ashworth Scale> a 1+ in the elbow and wrist flexors.
* Maintain seated position without human support or assistance for at least 10 seconds and maintain standing position for more than 30 seconds to perform transfers from one surface to another.

Exclusion Criteria:

* Altered cognitive ability, assessed through the "Short Portable Mental State Questionnaire".
* Application of botulinum toxin within six (6) months prior to participation in the study.
* Patients with skin lesions, lacerations or allergies.
* People with pacemaker.
* People in whom the H reflex can not be evoked.
* Pain and hyperalgesia in the upper limb.
* Peripheral vascular disease in upper limb.
* Fractures, or musculoskeletal injuries in the paretic upper limb less than a year old.
* Osteoarthritis, rheumatoid arthritis and clinical conditions associated with acute pain, inflammation, and moderate to severe decrease in joint mobility.
* Consumption of drugs such as Baclofen, benzodiazepines, or muscle relaxants such as dantrolene and tizanidine.
* Ingestion of caffeine and alcohol 12 hours before evaluations.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-24 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Muscular tone of wrist and elbow flexors. | before (baseline) and immediately after the intervention (maximum 10 minutes after the intervention).
  Defined as the resistance to movement of passive movement, it will be evaluated by the Modified Ashworth Scale (EAM) in flexo-extensors of the elbow and wrist and hand. (Ordinal scale of 6 points, with a range from 0 = normal tone to 4 = rigid segment in flexion or extension) .109 The EAM includes an additional degree of 1+, which has a sub-classification between an increase level and an increase of speed in the tone.
Reflex excitability of the flexor carpi radialis. | before (baseline) and immediately after the intervention (maximum 10 minutes after the intervention).
  Excitability is a specific property of muscle and nerve tissue and occurs when depolarization exceeds the threshold level in the action potential. The excitability will be measured from the evocation of H Reflex in the flexor carpi radialis muscle (FRC).
Joint kinematics in Functional Reach Pattern | before (baseline) and immediately after the intervention (maximum 10 minutes after the intervention).
  Shoulder, elbow and trunk angles (degrees), trunk displacement (cm) and duration (sec) of the Functional Reach Pattern (PAF) will be evaluated with the software Contemplas.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Juliana González Silva, Principal Investigator — Universidad Industrial de Santander

IPD SHARING:
Plan to Share IPD: No
It is not contended to share the data.